CLINICAL TRIAL: NCT01318356
Title: The Qure Study: Q-fever Fatigue Syndrome - Response to Treatment
Acronym: Qure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Stephan Keijmel, S.P. Keijmel, MD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205520003-20110307; 2011-000643-25 (EudraCT Number)
Record Dates: First submitted 2011-03-15; First posted 2011-03-18 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Q Fever; Fatigue Syndrome, Chronic; Coxiella Infection
Keywords: Q fever; Cognitive behavioral therapy; Doxycycline; Fatigue; Coxiella
MeSH Terms: conditions — Q Fever; Fatigue Syndrome, Chronic; Fatigue | interventions — Cognitive Behavioral Therapy; Doxycycline; Tetracycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy
- Doxycycline (Experimental)
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — CBT will consist of a protocolized intervention of 12 sessions during a period of 24 weeks. It starts with goal setting and psycho-education on the possible role of cognitions and behavior in maintaining the fatigue. The maintaining factors will subsequently be addressed (regulation of sleep-wake cycle, gradual increasing activity, reformulating fatigue related cognitions).
  Other Names: Behavior Therapy, Cognitive; Cognition Therapy; Cognitive Behavior Therapy; Cognitive Psychotherapy; Psychotherapy, Cognitive; Therapy, Cognition; Therapy, Cognitive; Therapy, Cognitive Behavior
  Arms: Cognitive behavioral therapy
Drug: Doxycycline — Antibiotic therapy will consist of doxycycline once daily 200 mg (in 1 capsule) for 24 weeks. Patients will be monitored 4, 8, 16 and 26 weeks after start for side effects (rash, liver enzymes). Antibiotics will be stopped in case of side effects or pregnancy.
  Other Names: Doxycycline Monohydrate; Tetracycline
  Arms: Doxycycline
Drug: Placebo — Patients in the placebo group will receive once daily 1 placebo capsule identical in appearance to the doxycycline for 24 weeks and have the same visits and monitoring for side effects as the patients randomized to doxycycline (Patients will be monitored 4, 8, 16 and 26 weeks)
  Other Names: Sham Treatment
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the efficacy of two treatment strategies for fatigue and disabilities in QFS: long term treatment with doxycycline or cognitive behavioral therapy (CBT).

DETAILED DESCRIPTION:
Q fever fatigue syndrome (QFS) is one of the most frequent sequelae of Q fever, and constitutes a significant problem in the current outbreak of Q fever. QFS leads to substantial morbidity and has a high socio-economic burden, related to increased use of healthcare facilities and absence from work. It is envisaged that over 750 patients will become chronically fatigued due to Q fever in The Netherlands (20% of 4000 patients from 2007 until now). Although the outbreak appears to diminish, it is expected that Q fever will remain an endemic disease, and therefore this number will continue to grow. A vast medical consumption can be anticipated, stressing the need for an accessible and effective intervention and clear treatment guidelines.

The study will contribute to a better understanding of effective treatment of QFS, providing evidence-based guidelines for general practitioners and medical specialists.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-lactating females who are 18 years or older
* Laboratory-proven acute Q fever since the year 2007 and/or positive serology fitting a past infection with Coxiella burnetii;
* AND being severely fatigued, defined by scoring 35 or higher on the subscale fatigue severity of the CIS;
* AND being fatigued for at least 6 months;
* AND disabled because of the fatigue, defined by scoring 450 or higher on the SIP
* Subjects must sign a written informed consent form.

Exclusion Criteria:

* Fulfilling criteria for chronic Q fever, namely:

  * IFA IgG fase I ≥ 1024, ≥ 3 months after acute Q fever and/or
  * Positive Coxiella burnetii PCR on serum or tissue, 1 month after acute Q fever
* Acute Q fever in the setting of a prosthetic cardiac valve or aneurysm surgery or stenting necessitating prophylactic use of doxycycline;
* Pregnancy or unwillingness to use effective contraceptives during the entire study period;
* Imminent death;
* Inability to give informed consent;
* Allergy or intolerance to doxycycline;
* Somatic or psychiatric illness that could explain the chronic fatigue;
* Subjects who are currently enrolled on other investigational drug trials or receiving investigational agents;
* Receiving antibiotics for more than 4 weeks, potentially active against Coxiella burnetii, for any other reason since Q-fever diagnosis;
* Subjects who are receiving and cannot discontinue barbiturates, phenytoin, or carbamazepine (these drugs may increase the metabolism of doxycycline and therefore reducing half-life of doxycycline);
* Moderate or severe liver disease (AF, ALAT, ASAT > 3 times the upper limit of normal).
* Current engagement in a legal procedure concerning financial benefits (only current involvement interferes with the effectivity of cognitive behavioral therapy. Once the appeal procedure ends, subjects can be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chantal P Bleeker-Rovers, MD PhD, Study Director — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Keijmel SP, Delsing CE, Sprong T, Bleijenberg G, van der Meer JW, Knoop H, Bleeker-Rovers CP. The Qure study: Q fever fatigue syndrome--response to treatment; a randomized placebo-controlled trial. BMC Infect Dis. 2013 Mar 27;13:157. doi: 10.1186/1471-2334-13-157. PMID 23536997
- [Derived] Keijmel SP, Delsing CE, Bleijenberg G, van der Meer JWM, Donders RT, Leclercq M, Kampschreur LM, van den Berg M, Sprong T, Nabuurs-Franssen MH, Knoop H, Bleeker-Rovers CP. Effectiveness of Long-term Doxycycline Treatment and Cognitive-Behavioral Therapy on Fatigue Severity in Patients with Q Fever Fatigue Syndrome (Qure Study): A Randomized Controlled Trial. Clin Infect Dis. 2017 Apr 15;64(8):998-1005. doi: 10.1093/cid/cix013. PMID 28329131

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 156 patients signed informed consent and were randomized; of these, 155 started treatment, either doxycycline (n = 52), placebo (n = 52), or CBT (n = 51). One patient refused double-blind randomization after allocation to the medication group, and received no treatment.
Groups:
- Cognitive Behavioral Therapy: Cognitive behavioral therapy: CBT will consist of a protocolized intervention during a period of 24 weeks. It starts with goal setting and psycho-education on the possible role of cognitions and behavior in maintaining the fatigue. The maintaining factors will subsequently be addressed (regulation of sleep-wake cycle, gradual increasing activity, reformulating fatigue related cognitions).
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy | Doxycycline | Placebo
Started | 51 | 52 | 52
Completed | 43 | 49 | 50
Not Completed | 8 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy | Doxycycline | Placebo | Total
Number analyzed (Participants) | 51 | 52 | 52 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.7) | 43.6 (10.2) | 44.6 (12.3) | 43.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 20 | 74
  Male | 26 | 23 | 32 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 51 | 52 | 52 | 155
Sickness Impact Profile 8 total score [Mean (Standard Deviation); unit: scores on a scale] — The SIP is an instrument that is used to gauge sickness-related dysfunction. The weighted total score on eight subscales of the SIP8 (SIP8 total score) will be used to assess functional disability in all domains of functioning. Values range from 0-4999. Higher scores reflect a higher level of functional impairment.
  scores on a scale | 1369.4 (646.7) | 1304.9 (537.7) | 1295.1 (593.7) | 1322.8 (591.1)
Checklist Individual Strength, subscale fatigue [Mean (Standard Deviation); unit: scores on a scale] — The primary outcome measure is the fatigue severity measured by the subscale fatigue severity (8 items, 7-point Likert Scale) of the Checklist Individual Strength (CIS questionnaire) with a severity range from 8-56. High scores indicate a high level of fatigue. Patients with a cut-off score of ≥35 are classified as severely fatigued.
  scores on a scale | 49.7 (4.7) | 51.4 (4.7) | 50.2 (4.8) | 50.36 (4.9)
Symptom Checklist 90 total score [Mean (Standard Deviation); unit: scores on a scale] — Level of psychological distress measured with the total score of the Symptom Checklist 90 (SCL90). The SCL90 consist of 90 items scored on a fivepoint scale. Scores range from 90-450. A low total score reflects psychological well-being.
  scores on a scale | 156.4 (35.0) | 152.2 (31.4) | 159.1 (41.0) | 155.6 (36.0)
Duration of symptoms [Median (Inter-Quartile Range); unit: months] | 40 [22 to 59] | 36 [24.25 to 57] | 37.50 [25.50 to 50.75] | 39 [24 to 54]

OUTCOME MEASURES:

1. Primary Outcome: Checklist Individual Strength (CIS)
Description: The primary outcome measure is the fatigue severity measured by the subscale fatigue severity (8 items, 7-point Likert Scale) of the Checklist Individual Strength (CIS questionnaire) with a severity range from 8-56. High scores indicate a high level of fatigue. Patients with a cut-off score of ≥35 are classified as severely fatigued.
Time Frame: 24 weeks after start of treatment
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Doxycycline | Placebo
Number analyzed (Participants) | 50 | 52 | 52
score on a scale | 31.6 [28.0 to 35.1] | 40.8 [37.3 to 44.3] | 37.8 [34.3 to 41.2]

2. Secondary Outcome: Sickness Impact Profile (SIP) Total Score
Description: Level of functional impairment measured with the Sickness Impact Profile (SIP). The SIP is an instrument that is used to gauge sickness-related dysfunction. The weighted total score on eight subscales of the SIP8 (SIP8 total score) will be used to assess functional disability in all domains of functioning (range 0-5799). A higher score indicates higher levels of functional impairment. A score of 450 or higher on the SIP is defined as being significant disabled because of fatigue.
Time Frame: 24 weeks after start of treatment
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Doxycycline | Placebo
Number analyzed (Participants) | 50 | 52 | 52
score on a scale | 786.8 [615.3 to 958.3] | 1101.5 [933.5 to 1269.6] | 963.8 [795.8 to 1131.9]

3. Secondary Outcome: Symptom Checklist 90 (SCL90)
Description: The total score of the Symptom Checklist 90 (SCL90) measures the level of psychological distress. The SCL90 consists of 90 items scored on a 5-point scale. Scores range from 90 to 450. A low total score reflects high psychological well-being. The SCL-90 is a reliable and valid instrument.
Time Frame: 24 weeks after start of treatment
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Doxycycline | Placebo
Number analyzed (Participants) | 50 | 52 | 52
score on a scale | 127.1 [119.4 to 134.7] | 149.2 [141.6 to 156.7] | 142.6 [134.1 to 150.1]

ADVERSE EVENTS:
Time Frame: Safety was assessed by monitoring adverse events (AEs) and concomitant drug use. For patients allocated to the medication condition, AEs were monitored at 4 weeks, 8 weeks, and 16 weeks after start of therapy, and at EOT (= up to approximately 26 weeks after start of therapy). Furthormore, if applicable, during the trial when reported by the patient. For patients allocated to CBT, AEs were monitored at 8 weeks after start of therapy, and at EOT (up to 26 weeks after start of therapy).
Arm/Group | Cognitive Behavioral Therapy | Doxycycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52 | 2/52
Other Adverse Events (participants affected / at risk) | 42/50 | 51/52 | 45/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioral Therapy (N=50) | Doxycycline (N=52) | Placebo (N=52)
Urosepsis (Renal and urinary disorders) | 0 | 0 | 1 — One patient who had not yet started treatment was admitted to hospital with urosepsis.
Cardiological symptoms (Cardiac disorders) | 0 | 0 | 1 — The other patient was admitted for clinical evaluation of preexisting cardiological symptoms, which yielded no diagnosis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (N=50) | Doxycycline (N=52) | Placebo (N=52)
Infection (Infections and infestations) | 29 (54) | 22 (33) | 26 (46)
Gastointestinal (Gastrointestinal disorders) | 5 (5) | 31 (51) | 27 (33)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 14 (18) | 22 (28) | 17 (22)
Skin (Skin and subcutaneous tissue disorders) | 5 (5) | 20 (29) | 10 (12)
Neurological (Nervous system disorders) | 6 (8) | 13 (13) | 10 (11)
Bone and teeth (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 2 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0)
Other (General disorders) | 18 (21) | 24 (34) | 13 (15)
Laboratorial (Investigations) | 0 (0) | 14 (16) | 7 (8)

LIMITATIONS AND CAVEATS:
It was not designed to compare doxycycline and CBT directly, due to the limited number of available patients.

As masking for CBT was not possible, this trial was partly blinded. CBT was directly compared to placebo plus usual care.

Due to the maximum number of vailable patients, it was not possible to include a control group without any form of treatment.

Finally, it is unclear whether the detected effects will be sustained over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No